CLINICAL TRIAL: NCT03332862
Title: Acute Efficacy of Point-by-point Radiofrequency Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation: a Randomized Comparison of Continuous Versus Discontinuous Design of Encircling Lesions
Brief Title: Continuous Versus Discontinuous Design of Encircling Lesions During Ablation for Atrial Fibrillation
Acronym: CDAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Charles University, Czech Republic (Other); 3rd Department of Internal Medicine - Cardiology (Unknown)
Responsible Party: Principal Investigator, Bashar Aldhoon, Dr. Bashar Aldhoon, PhD, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-17-06-22
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation; Atrial Fibrillation; Contact Force; Continuous Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuous ablation (Experimental): perform discontinuous ablation of ipsilateral pulmunary veins.
  Interventions: Procedure: catheter ablation
- Continuous ablation (Active Comparator): perform continuous ablation of ipsilateral pulmunary veins.
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — catheter ablation for atrial fibrillation treatment

SUMMARY:
Acute efficacy of point-by-point radiofrequency ablation for pulmonary vein isolation in patients with atrial fibrillation are comparable independantly of the ablation strategy (continous versus discontinuous ablation) under the same condition of power delivery.

DETAILED DESCRIPTION:
The number of pulmonary vein isolation (PVI) therapy for atrial fibrillation (AF) is increasing. Durable PVI is cornerstone for long-term freedom of AF. In one previous study continuous ablation was suggested to be more efficient in durable PVI. However, this hypothesis has not been proven in randomized fashion.

The current study is to confirm whether continuous versus discontinuous design of encircling lesions are comparable under the same conditions of power delivery.

The study design is a two-centre prospective randomized trial to compare the acute efficacy by using the above described approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pulmonary vein isolation with radiofrequency catheter ablation for paroxysmal atrial fibrillation treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Combined unsuccessful PVI or PV reconnection | 30 min after ablation
  Combined unsuccessfuk PVI after completeing the primary lesion set or PV reconnection during the waiting time

SECONDARY OUTCOMES:
Early pulmunary veins reconnection | 10 min.
  Early pulmunary veins reconnection within the first 10 min after PVI

CONTACTS AND LOCATIONS:
Overall Officials: Bashar Aldhoon, MD, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Aldhoon B, Peichl P, Osmancik P, Konecny P, Kautzner J, Wichterle D. Acute efficacy of contiguous versus temporally discontiguous point-by-point radiofrequency pulmonary vein isolation in patients with paroxysmal atrial fibrillation: a randomized study. J Interv Card Electrophysiol. 2022 Sep;64(3):661-667. doi: 10.1007/s10840-021-01113-9. Epub 2022 Jan 6. PMID 34988847